CLINICAL TRIAL: NCT01805791
Title: A Phase III, Randomized, Multi-Centre, Double-Blind, Placebo-Controlled Trial of HMPL-004 in Patients With Mild to Moderate Active Ulcerative Colitis
Brief Title: A Phase III Trial of HMPL-004 in Patients With Mild to Moderate Active Ulcerative Colitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim futility analysis results
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMPL-004-03
Record Dates: First submitted 2013-03-04; First posted 2013-03-06 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2018-07

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis,; UC; Patients; active; mild; moderate
MeSH Terms: conditions — Colitis, Ulcerative; Motor Activity; Lymphoma, Follicular | interventions — Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were randomized according to a stratified blocked randomization schedule generated by an unblinded biostatistician. Stratification was by country/region and modified Mayo Score at screening using an interactive web-based response system (IWRS).

ARMS (3):
- Placebo (Placebo Comparator): Placebo, oral tablets, three times a day
  Interventions: Drug: Placebo
- HMPL-004 1800 mg/day (Experimental): 1 600 mg HMPL-004 tablet, 2x400 mg placebo tablets taken 3 times a day
  Interventions: Drug: HMPL-004 1800 mg/day
- HMPL-004 2400 mg/day (Experimental): 2 x 400 mg HMPL tablets, 1 x 600 mg placebo tablet, taken 3 times per day
  Interventions: Drug: HMPL-004 2400 mg/day

INTERVENTIONS:
Drug: HMPL-004 1800 mg/day — Subjects randomized to the arm of HMPL-004 1800 mg/day will receive HMPL-004 600 mg TID (total dose 1800 mg/day) for 56 days (8 weeks).
  Other Names: Chuan xinlian
  Arms: HMPL-004 1800 mg/day
Drug: Placebo — Subjects randomized to the arm of Placebo will receive matching Placebo three times daily for 56 days (8 weeks).
  Arms: Placebo
Drug: HMPL-004 2400 mg/day — Subjects randomized to the arm of HMPL-004 2400 mg/day will receive HMPL-004 800 mg TID (total dose 2400 mg/day) for 56 days (8 weeks).
  Other Names: Chuan xinlian
  Arms: HMPL-004 2400 mg/day

SUMMARY:
A placebo controlled study of two doses of HMPL-004 in patients with active mild to moderate ulcerative colitis (UC), with a modified Mayo Score 4-10 and an endoscopy subscore of 2-3, taking mesalamine (or equivalent) as a concomitant medication.

The objective is to evaluate the efficacy and safety of HMPL-004 with mesalamine (mesalamine treatment failures). Efficacy will be measured by a comparison of the proportion of patients in each treatment group attaining clinical remission at Week 8 as compared to placebo.

DETAILED DESCRIPTION:
This Phase III study of HMPL-004 was to enroll approximately 420 subjects with active mild to moderate ulcerative colitis (UC; modified Mayo Score 4-10 and endoscopy score of 2-3). The trial included male and female subjects aged 18 or older. Subjects were currently receiving ≥2.4 g/day mesalamine or equivalent, provided they had taken 5-aminosalicylate (ASA; i.e., mesalamine) at a dose ≥2.4 g/day for at least 6 weeks prior to randomization and were on a stable dosage for at least 2 weeks prior to entering the screening phase of the study.

Qualifying subjects who entered into this study received 3 daily doses of oral HMPL 004 tablets or placebo for 56 days (8 weeks). There were 3 arms in this study consisting of placebo, HMPL-004 600 mg three times a day (TID) or 800 mg TID. Approximately 420 subjects were to be randomized 1:1:1 to one of these 3 arms, stratified by country/region in up to 150 clinical centers in North America, Europe, and Asia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be currently receiving mesalamine ≥ 2.4 g/day (or the equivalent) for at least 6 weeks prior to randomization and on a stable dosage for at least 2 weeks prior to entering the screening phase of the study to ensure a stable dose is established at least 2 weeks prior to the endoscopic procedures.
* Have active mild to moderate ulcerative colitis defined by a modified Mayo Score 4-10, and with endoscopy score activity of 2-3 points confirmed by centrally read colonoscopy (within 2 weeks prior to randomization.
* Minimum modified Mayo endoscopy score of >2 at the time of study colonoscopy.
* Age ≥ 18 years.
* Patients have no prior exposure to HMPL-004.
* Have adequate renal, hepatic and bone marrow function (see exclusion criteria).
* All fertile male and female subjects must agree to use one of the following types of contraception: abstinence, intrauterine device, implantable progesterone device, and progesterone intramuscular injection, oral contraceptive which has been started at least one month prior to visit one and continues for the duration of the trial, contraceptive patch, or condom with spermicide.
* Show evidence of a personally signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial

Exclusion Criteria:

1. Subjects with intolerance or adverse reactions to mesalamine (or equivalent medications).
2. Diagnosed with Crohn's Disease or with lesions such as fistulas or granulomas on biopsy noted either in history or at baseline endoscope, which would be suspicious for Crohn's disease, or with a diagnosis of indeterminate colitis. Subjects with Primary Sclerosing Cholangitis (PSC) are excluded..
3. Severe disease with an ulcerative colitis modified Mayo Clinic score above 10 points at baseline.
4. Positive stool test for pathogens for sample taken within the previous 2 weeks prior to study entry.
5. Active Clostridium difficile (C. diff) infection.
6. Use of Inflammatory Bowel Disease related herbal supplements including but not limited to supplements containing andrographis and probiotics two weeks prior to study entry or during the study.
7. Toxic megacolon or toxic colitis.
8. Probable requirement for intestinal surgery within 12 weeks after the start of study medication.
9. Receiving oral or rectal steroids within 1 month prior to study entry.
10. Receiving rectal mesalamine within one week prior to study entry.
11. Receiving azathioprine, 6-mercaptopurine, methotrexate, tacrolimus, cyclosporine, or other immunosuppressive therapy at the time of screening or within the preceding 6 weeks.
12. Receiving anti-tumor necrosis factor-α agents such as infliximab, adalimumab, golimumab, or certolizumab pegol at the time of screening or within the preceding 8 weeks.
13. Receiving other investigational drugs or biologics within 1 month or five half lives.
14. Receiving antibiotics within 2 weeks of study entry.
15. Hemoglobin concentration < 9 g/dl.
16. White blood cell count (WBC) below 3,000/cmm, or platelets below 100,000/cmm.
17. Serum glutamate oxaloacetate transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT), alkaline phosphatase >2.5 upper limit of normal.
18. Serum creatinine >1.5 times upper limit of normal.
19. Significant concurrent medical diseases including: active peptic ulcer disease; uncompensated congestive heart disease; myocardial infarction within the last 12 months; unstable angina pectoris; uncontrolled hypertension; pulmonary disease requiring oxygen therapy.
20. Chronic Hepatitis B or any history of Hepatitis C.
21. Previous colonic surgery except for simple polypectomy or appendectomy. .
22. History of cancer within the last 5 years other than resected cutaneous basal and squamous cell carcinomas, and in situ cervical cancer.
23. Patients with a history of or concurrent colonic dysplasia associated with UC, except those with completely excised sporadic colorectal polyps.
24. Women who are pregnant or breast feeding.
25. Patients known to be seropositive for HIV, or who have had an AIDS defining illness, or a known immunodeficiency disorder.
26. Patients with a history of tuberculosis or exposure to tuberculosis, or a history of a chest X-ray suspicious for tuberculosis, unless confirmed to be purified protein derivative (PPD) skin test negative or latent tuberculosis that has been previously treated.
27. History of alcohol or drug abuse that would interfere with the ability to be compliant with the study procedure.
28. Known allergy to plants of the Acanthaceae family.
29. Unwillingness to participate in the study.
30. Any underlying medical condition that in the Investigator's opinion will make the administration of study drug hazardous to the patient or would obscure the interpretation of adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rongjun Liu, MD, Study Director — Hutchison Medipharma Limited
Locations (1):
- Clinical Research Management, Inc, Agawam, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HMPL-004 1800 mg/Day: 1 600 mg HMPL-004 tablet, 2x400 mg placebo tablets taken 3 times a day
  HMPL-004 1800 mg/day: Subjects randomized to the arm of HMPL-004 1800 mg/day will receive HMPL-004 600 mg 3 times daily (total dose 1800 mg/day) for 56 days (8 weeks).
- HMPL-004 2400 mg/Day: 2 x 400 mg HMPL tablets, 1 x 600 mg placebo tablet, taken 3 times per day
  HMPL-004 2400 mg/day: Subjects randomized to the arm of HMPL-004 2400 mg/day will receive HMPL-004 800 mg 3 times daily (total dose 2400 mg/day) for 56 days (8 weeks).
Period: Overall Study
Arm/Group | Placebo | HMPL-004 1800 mg/Day | HMPL-004 2400 mg/Day
Started | 66 | 67 | 68
Completed | 44 | 50 | 48
Not Completed | 22 | 17 | 20

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics are summarized in the Safety Population, by treatment.
Groups:
- Placebo: Placebo, oral tablets, 3 times a day
  Placebo: Subjects randomized to the arm of Placebo will receive matching Placebo three times daily for 56 days (8 weeks).
- HMPL-004 1800 mg/Day: 1 600 mg HMPL-004 tablet, 2x400 mg placebo tablets taken 3 times a day
  HMPL-004 1800 mg/day: Subjects randomized to the arm of HMPL-004 1800 mg/day will receive HMPL-004 600 mg 3 times a day (total dose 1800 mg/day) for 56 days (8 weeks).
- HMPL-004 2400 mg/Day: 2 x 400 mg HMPL tablets, 1 x 600 mg placebo tablet, taken 3 times a day
  HMPL-004 2400 mg/day: Subjects randomized to the arm of HMPL-004 2400 mg/day will receive HMPL-004 800 mg 3 times a day (total dose 2400 mg/day) for 56 days (8 weeks).
- Total: Total of all reporting groups
Arm/Group | Placebo | HMPL-004 1800 mg/Day | HMPL-004 2400 mg/Day | Total
Number analyzed (Participants) | 66 | 67 | 68 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (16.32) | 43.9 (15.07) | 40.6 (12.33) | 43.2 (14.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 37 | 33 | 93
  Male | 43 | 30 | 35 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 10 | 28
  Not Hispanic or Latino | 57 | 58 | 58 | 173
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 9 | 14
  White | 62 | 63 | 55 | 180
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4
Current Smoker: Yes, No [Count of Participants; unit: Participants]
  Yes | 6 | 4 | 1 | 11
  No | 60 | 63 | 67 | 190
Weight, Continuous [Mean (Standard Deviation); unit: kg] | 80.94 (16.00) | 79.77 (19.35) | 82.24 (21.42) | 80.99 (19.01)
Height, Continuous [Mean (Standard Deviation); unit: cm] | 172.21 (10.30) | 170.67 (9.54) | 170.28 (8.74) | 171.05 (9.53)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a Clinical Remission at Week 8
Description: Clinical remission was defined as a total Mayo Score of ≤2 points with no individual sub-score >1 point and rectal bleeding score = 0.
Time Frame: 8 weeks
Population: Analysis included only those subjects who were randomized on or prior to 16 Jun 2014 and had an opportunity to complete the 8 week treatment period. Worst case imputation imputed any missing Week 8 value as a failure.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo, oral tablets, 3 times a day
  Placebo: Subjects randomized to the arm of Placebo will receive matching Placebo 3 times a day for 56 days (8 weeks).
Arm/Group | HMPL-004 2400 mg/Day | HMPL-004 1800 mg/Day | Placebo
Number analyzed (Participants) | 57 | 58 | 52
Participants | 9 | 7 | 9

2. Secondary Outcome: The Proportion of Subjects With Clinical Response at Week 8
Description: Clinical response was defined as a decrease in a modified Mayo Score from baseline by ≥3 points and ≥30% decrease in the modified Mayo Score, along with either a decrease in the rectal bleeding score ≥1 or an absolute rectal bleeding score ≤1.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 2400 mg/Day | HMPL-004 1800 mg/Day | Placebo
Number analyzed (Participants) | 57 | 58 | 52
Participants | 23 | 19 | 16

3. Secondary Outcome: The Proportion of Subjects With Mucosal Healing at Week 8
Description: Mucosal healing was defined as having normal or inactive disease using a modified Mayo Score to determine if the decrease in the modified Mayo endoscopy sub-score from baseline was ≥1 in at least 1 segment and had an absolute score ≤1 in all segments.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 2400 mg/Day | HMPL-004 1800 mg/Day | Placebo
Number analyzed (Participants) | 57 | 58 | 52
Participants | 13 | 13 | 14

ADVERSE EVENTS:
Time Frame: 86 days
Arm/Group | HMPL-004 2400 mg/Day | HMPL-004 1800 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/67 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67 | 4/66
Other Adverse Events (participants affected / at risk) | 31/68 | 25/67 | 21/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HMPL-004 2400 mg/Day (N=68) | HMPL-004 1800 mg/Day (N=67) | Placebo (N=66)
Pyrexia (General disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HMPL-004 2400 mg/Day (N=68) | HMPL-004 1800 mg/Day (N=67) | Placebo (N=66)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 1
GERD (Gastrointestinal disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No